CLINICAL TRIAL: NCT06686095
Title: Comparison of Analgesic Effect of Adductor Canal Block, IPACK, and Genicular Nerve Block Following Total Knee Arthroplasty Under Spinal Anesthesia
Brief Title: Analgesic Effect of Adductor Canal Block, IPACK Block, and Genicular Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Selcuk KAYIR, Associate Professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-81
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Adductor Canal Block; Ipack block; Genicular nerve block; Post-Operative Pain; Peripheral Nerve Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group A (n=30): Patients who underwent adductor canal block , group I (n=30): Patients who underwent infiltration block between popliteal artery and knee capsule block, group G (n=30): Patients who underwentgenicular nerve block
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Adductor canal block (Active Comparator): Patients who underwent adductor canal block
  Interventions: Procedure: Group Adductor canal block
- Group IPACK Block (Active Comparator): Patients who underwent Infiltration between Popliteal Artery and Capsule of the Knee block
  Interventions: Procedure: Group IPACK Block
- Group Genicular Nerve Block (Active Comparator): Patients who underwent Genicular nerve block
  Interventions: Procedure: Group Genicular Nerve Block

INTERVENTIONS:
Procedure: Group Adductor canal block — Adductor canal block procedure: The patient will be informed about the technique and consent will be obtained. The patient's hip will be slightly externally rotated, and an ultrasonography linear probe will be placed on the medial thigh, at the midpoint of the patella and vastus medialis. After locating the femoral artery at approximately 3-4 cm depth, if not visible, the artery can be traced distally from the inguinal region using Doppler mode. Once the vastus medialis and sartorius muscles are identified, the superficial femoral artery is centered at the midpoint of the sartorius muscle. The adductor canal roof, along with the saphenous and vastus medialis nerves, appears as hyperechoic structures. A needle is inserted in-plane, advancing toward the anterolateral femoral artery aspect, and 5-20 mL of LA is injected.
  Arms: Group Adductor canal block
Procedure: Group Genicular Nerve Block — Genicular Nerve Block: The patient is informed and consent is obtained. With a pillow in the popliteal fossa, the knee is slightly flexed. For the superior lateral genicular nerve, a linear USG probe is positioned on the lateral femoral epicondyle, moving proximally to visualize the bone metaphysis. The superolateral artery is seen between the vastus lateralis fascia and the femur. Using in-plane or out-of-plane technique, the needle is guided to the bone, and 4-5 mL of LA is injected. For the superior medial nerve, the probe is placed on the medial epicondyle and moved proximally to visualize the bone near the adductor tubercle. The artery lies between the femur and vastus medialis fascia. For the inferomedial artery, the probe is placed on the tibial medial condyle, moving distally. A negative aspiration test is conducted before each LA injection.
  Arms: Group Genicular Nerve Block
Procedure: Group IPACK Block — IPACK Block: Before the procedure, the patient is informed about the technique and written consent is obtained from the patient. The patient lies in the prone position. The linear USG probe is placed approximately 2-3 cm above the popliteal fossa and scanned distally to identify the femoral shaft and popliteal artery. If the femoral condyles are initially visualized, the probe is moved until the condyles disappear and the femoral shaft is identified as a straight line and hyperechoic. Color doppler can be used to identify the popliteal vessels. The peripheral block needle is advanced between the femoral shaft and the popliteal artery. After negative aspiration control, 15-20 mL of LA medication is injected here.
  Arms: Group IPACK Block

SUMMARY:
Patients with total knee arthroplasty (TKA) experience severe postoperative pain. This reduces patient satisfaction, delays mobility, and prolongs hospital stay. Peripheral nerve blocks, which are part of multimodal analgesia, are widely used in postoperative pain management. In this study, the effects of adductor canal block (ACB), popliteal artery and knee capsule infiltration block (IPACK), and genicular nerve block (GSB) on postoperative VAS score, opioid consumption, and mobility were investigated.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a surgical procedure performed on patients with severe pain and severely limited range of motion in the knee joint due to knee osteoarthritis, when traditional conservative treatments have failed. Fifty-eight percent of patients who undergo TKA experience moderate or severe pain in the postoperative period. Inadequate pain control leads to complications such as venous thrombosis, coronary ischemia, myocardial infarction, and pneumonia, and increases morbidity. In addition, failure to control postoperative pain negatively affects physical therapy procedures. This situation prolongs the rehabilitation and hospital stay of patients, thus increasing care costs. Therefore, it is of great importance to reduce the patient's pain after TKA.

Femoral nerve block (FNB) has traditionally been a critical component of multimodal analgesia in TKA due to its high analgesic efficacy. However, FNB limits physical therapy by causing motor limitations in the quadriceps muscle. This situation causes delays in ambulation and discharge. Due to the difficulties in rehabilitation observed in patients undergoing FNB due to quadriceps muscle weakness, different techniques were sought and the Adductor canal block (ACB) emerged. AKB is a sensory block that blocks the saphenous nerve, a sensory nerve that courses in the adductor canal in the thigh, thus preserving motor function. It is an alternative block to FNB by providing adequate analgesia to the anterior compartment of the knee.

Genicular nerves include branches of the femoral, common peroneal, saphenous, tibial and obturator nerves that innervate the knee capsule. It is known that the superolateral, superomedial and inferomedial branches of the genicular nerve are close to the periosteum of the tibia and femur and play a role in sensory innervation of the anterior part of the knee joint. Genicular nerve block (GNB) is used in chronic osteoarthritis pain and has been used in recent years to relieve postoperative pain in TKA.

Infiltration between Popliteal Artery and Capsule of the Knee (IPACK block) is performed by infiltrating local anesthetic (LA) between the popliteal artery and the knee capsule under USG guidance. The sciatic nerve has an important function in the motor and sensory innervation of the posterior leg. In the IPACK block application, the LA spreads along the popliteal fossa and proximal sciatic nerve involvement does not occur. Thus, the sensory nerve network innervating the posterior part of the knee is blocked. Since IPACK block provides only sensory block without causing motor block, it is a new method recommended for analgesia in knee surgery as an alternative to sciatic nerve block, which causes motor block.

Method:

Exclusion criteria from the study were: patient refusal to participate in the study, patients with ASA physical classification 4-5, revision TKA, simultaneous bilateral TKA, patients younger than 18 years and older than 80 years, BMI >40, allergy to the local anesthetic used, DM, hepatic and renal failure, alcohol and drug addiction, high-dose opioid drug use within 3 days before surgery, peripheral nerve disease, patients who could not score pain with the VAS system, patients with contraindications to spinal anesthesia and peripheral nerve block.

Adductor canal block procesure: Before the procedure, the patient will be informed about the technique and a signed consent will be obtained from the patient. The patient's hip will be slightly externally rotated and the ultrasonography linear probe will be placed on the medial aspect of the thigh, at the midpoint of the patella and vastus medialis. After the femoral artery is visualized at a depth of approximately 3-4 centimeters (cm) from the distal short axis angle, if the artery cannot be identified, the femoral artery, which is visualized in the inguinal region, can be followed distally starting from the proximal and the pulsatile flow of the artery will be seen in the doppler mode. After the vastus medialis and sartorius muscles are visualized, the superficial femoral artery is centered at the midpoint of the sartorius muscle. At this point, the roof of the adductor canal can be visualized. After the saphenous nerve and vastus medianus nerve are seen as small round hyperechoic structures, the needle is inserted with the in plane technique and advanced towards the anterolateral aspect of the superficial femoral artery. Then, 5-20 milliliters (mL) of LA is administered into the adductor canal.

Genicular Nerve Block: Before the procedure, the patient is informed about the technique and approval is obtained from the patient. A pillow is placed in the popliteal fossa of the patient lying in the supine position and the knee is slightly flexed. For superior lateral Genicular nerve blockade; the linear USG probe is placed on the lateral epicondyle of the femur in the coronal plane and moved proximally to visualize the metaphysis of the bone. At this level, the superolateral genicular artery can be seen between the deep fascia of the vastus lateralis and the femur. With the in-plane or out-of-plane technique, the peripheral block needle is advanced from the side of the artery until it touches the bone surface and 4-5 mL of LA medication is injected. For superior medial Genicular nerve blockade; the linear USG probe is placed on the medial epicondyle of the femur in the coronal direction and moved proximally to visualize the metaphysis of the bone in front of the adductor tubercle. The superior medial Genicular artery is seen between the femur and the deep fascia of the vastus medialis muscle. The peripheral block needle is inserted from the side of the artery until it touches the bone surface with an in-plane or out-of-plane technique and 4-5 ml of LA drug is injected. A linear USG probe placed coronally on the medial condyle of the tibia is moved distally to visualize the bone metaphysis. The inferomedial genicular artery can be seen under the medial collateral ligament. The peripheral block needle is inserted from the side of the artery until it touches the bone surface with an in-plane or out-of-plane technique and 4-5 ml of LA drug is injected. A negative aspiration test is performed before injecting LA drug in all blocks.

IPACK Block: Before the procedure, the patient is informed about the technique and written consent is obtained from the patient. The patient lies in the prone position. The linear USG probe is placed approximately 2-3 cm above the popliteal fossa and scanned distally to identify the femoral shaft and popliteal artery. If the femoral condyles are initially visualized, the probe is moved until the condyles disappear and the femoral shaft is identified as a straight line and hyperechoic. Color doppler can be used to identify the popliteal vessels. The peripheral block needle is advanced between the femoral shaft and the popliteal artery. After negative aspiration control, 15-20 mL of LA medication is injected here.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* BMI < 40
* 18-80 years old

Exclusion Criteria:

* ASA IV-V
* <18 years, >80 years
* Will undergo revision TKA surgery
* Will undergo bilateral TKA surgery
* BMI > 40
* Patients who used high dose opioid medication within 3 days before surgery
* those with widespread chronic pain, diabetes mellitus, a history of neuromuscular disease, hepatic and renal failure
* who underwent general anesthesia during the intraoperative period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Examination with Numeric Rating Scale | 48 hours
  Determination of patients' post-operative pain level. The Numeric Rating Scale (NRS), a method that converts the patient's pain perception into a numerical form, will be used to assess postoperative pain. NRS has a numerical scale ranging from 0 to 10. The patient will rate the intensity of pain on a scale from 0, indicating no pain, to 10, representing the worst imaginable pain (NRS 0=no pain, 4=mild to moderate pain, 6-8=severe pain, and >8=intolerable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Erol Olcok Training and Research Hospital, Çorum, Turkey (Türkiye)